CLINICAL TRIAL: NCT03418311
Title: Impact of Cervical Pessary Treatment for Prevention of Spontaneous Preterm Birth in Twin Pregnancies With Cervical Shortening on Children's Long-Term Survival Without Neurodevelopmental Disability: THE IMPETUS-TRIAL
Brief Title: Cervical Pessary Treatment for Prevention of s PTB in Twin Pregnancies on Children's Long-Term Outcome
Acronym: Impetus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bürgerhospital Frankfurt (Other)
Responsible Party: Principal Investigator, Ioannis Kyvernitakis, Associate Professor, Bürgerhospital Frankfurt
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BHFKIK2018I
Record Dates: First submitted 2018-01-23; First posted 2018-02-01 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-05

CONDITIONS: Preterm Birth; Premature Birth
Keywords: Twin pregnancy; Cervical Pessary; short cervix; Prevention
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control-Group (No Intervention): Control-group-women receive management as usual; i.e. expectant management with interventions only in terms of a tertiary prevention of PTB according to guidelines for premature rupture of membranes, premature labour or other pregnancy complications.
- Cervical Pessary-Group (Experimental): placement of the cervical pessary (non-invasive) at enrollment; removal of the cervical pessary (non-invasive) in a regular preventive examination at WoG 37.
  Interventions: Device: Cervical Pessary-Group

INTERVENTIONS:
Device: Cervical Pessary-Group — Placement of the cervical pessary (non-invasive) at enrolment including a transvaginal ultrasound to verify its correct fit. Removal of the cervical pessary (non-invasive) in a regular preventive examination at week of gestation 37+0. Except for placement/removal of cervical pessary the pregnant women will receive the usual care.
  Other Names: Arabin Cervical Pessary
  Arms: Cervical Pessary-Group

SUMMARY:
Preterm birth (PTB) complicates 13% of all pregnancies worldwide and is the most important cause of neonatal morbidity and mortality. Women with a twin pregnancy are at increased risk of preterm delivery. In the Netherlands, approximately 50% of women with a multiple pregnancy deliver before 37 weeks of gestation (WoG), of whom 9% deliver before 32 weeks. Evidence based treatment guidelines concerning prevention of PTB are not available in Europe. Expectant management is usual care with interventions only in terms of a tertiary prevention of PTB according to guidelines for premature rupture of membranes, premature labour or other pregnancy complications. The studies done on this topic included women at different stages of the second trimester so the question of the onset of cervix shortening and its impact on PTB is not answered yet. The critical period for a maximum impact of the pessary treatment on PTB is still to be verified. Up to now only the ProTwinTrial addressed the long-term outcome of the newborns, so here data and evidence is clearly missing. The investigators want to assess the impact of a cervical pessary treatment in twin pregnancies with cervical shortening on children's survival without neurodevelopmental disability at the age of 3 years at 3 different stages of the second trimester (16-20 (early) vs. 20-24 (middle) vs. 24-28 (late) weeks of gestation).

DETAILED DESCRIPTION:
Impetus is a prospective, multicentre, multinational, open-label, randomised, controlled clinical trail in parallel groups.

For sample size calculation, a the stratified design is accounted for and three equally large gestation groups assumed. For the pessary group a combined event rate of at least 8% for the primary outcome is assumed and for the comparison of the pessary group with the control group an odds ratio of 2.29 is assumed. This odds ratio correspond to the lower bound of a one-sided confidence interval for the event rate given in van´t Hooft (ProTwin Trial). To reach a power of at least 80%, at least 500 patients will be evaluated, 250 in the pessary group and 250 in the control group. To account for a drop out rate of 25%, overall n=672 pregnant women will be recruited.

The primary statistical aim is to compare the primary combined outcome "long-term survival without neuro-developmental disability at 3 years follow up" with a two-sided Cochran-Mantel-Haenszel-Test and a significance level of alpha=0.05. The primary outcome refers to a combined event in any of the twin and will be analysed for all pregnancies with available primary endpoint. The stratified study design is accounted by this stratified test according to the gestation groups.

The main statistical evaluation will be performed at two time points. (1) The complete data set for the secondary endpoints will be available after the last women enrolled in this study has delivered her twins, so the analysis of these outcome parameter will be done right after this event. (2) The primary outcome will be evaluated 3 years after the last woman enrolled in this study has delivered her twins. A descriptive analysis by preterm birth will be carried out calculating means and medians for quantitative variables and proportions with 95% confidence intervals for categorical variables. In general, statistical comparisons with the pessary arm and the control arms or other group comparisons for primary and secondary outcomes will be performed with stratified tests as well as comparisons in the gestation subgroups. Events will be analysed for each twin and for single children assuming appropriate random effect regression models. Further subgroup analyses regarding the cervical length will be performed (e.g. Cervical Length (CL) 15 to 25mm and below 15mm). All tests, see also examples in the synopsis, will be two-sided using a significance level of alpha=0.05.

For the primary endpoint a drop out rate of up to 25% is expected due to the long follow-up time (3 years) of the study; but no lost data for the secondary endpoints are expected because for these parameters the study has a short follow-up time till time to birth only.

An interim analysis shall be conducted on key safety parameters after birth of 300 twins: the following safety endpoints will be assessed by a one-sided test with alpha=1%

* on level of the neonates: rate of preterm birth, time to birth, birth weight, death, neonatal morbidity, harm of intervention
* and on the maternal level: rate of hospitalisation for threatened preterm labour < 32 weeks, rate of premature rupture of membranes (PRoM) <32 weeks, rate of infection / inflammation, rate of physical or psychological intolerance to pessary, rate of SAR/SAE, death.

The trial will be terminated as negative if a disadvantage for the pessary-treatment can be found in one of these tests. To guarantee a high safety level the significance level is chosen more conservatively than in a Bonferroni correction. All analysis will be carried out with SPSS® version 19.0 or later (IBM Company SPSS Inc. Headquarters, Chicago, Illinois. USA) and R version 3.2.3 or later (R Foundation for Statistical Computing, Vienna, Austria).

Methods against bias:

All women will be randomly allocated to the cervical pessary group or the control-group in a 1:1 ratio. The randomisation sequence is computer generated with variable block sizes using a web-based e-CRF (Online-Software Castor is a fully GCP compliant system) stratified for gestation groups and centers. The allocation code will be disclosed after the patient´s initials will be confirmed. The investigators or the trial coordinator will not have access to the randomization sequence.

Exclusion criteria were chosen to ensure an equal risk distribution for pregnancy complications and fetal morbidity / mortality rate for both study groups.

The study is open label since masking the intervention is not possible. All investigators should be trained in pessary application and cerclage placement. Quality protocols should be submitted according to the Clara-Angela Foundation requirements for pessary placement. Outcome assessors will be blinded to the interventions. Group allocations will base on an intention to treat basis with a per protocol allocation as sensitivity analysis.

The study will be registered and the study protocol is available. Outcome measures meet the core-outcome set for the evaluation of interventions to prevent PTB published by the crown-initiative in 2016.

ELIGIBILITY:
Inclusion Criteria:

* women with a diamniote twin pregnancy at 16-28 weeks of gestation with a shortened cervix ≤ 25 percentile
* women ≥ 18 years and capable of giving consent

Exclusion Criteria:

* monoamniote pregnancy
* major fetal abnormalities
* suspected twin-to-twin transfusion syndrome
* intrauterine death of one twin
* uterine malformation
* placenta previa totalis
* Cerclage prior to randomization
* active vaginal bleeding and/or spontaneous rupture of membranes and/or painful regular uterine contractions
* silicone allergy
* current participation in other RCT to avoid treatment conflicts

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — women being pregnant with a twin gestation
Enrollment: 672 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Children's survival without neurodevelopmental disability at the age of 3. | assesment of the newborns at age of 3 years (corrected age for prematurity)
  Recording of the mortality rate of the newborns; neurodevelopmental disability will be assessed by the Ages & Stages Questionnaire and by medical examination of the newborn at the age of 3 years

SECONDARY OUTCOMES:
rate of preterm birth | randomisation till birh, maximum 21 weeks
  rate of delivery before weeks of gestation 36+6 / 33+6 / 31+6 / 29+6 / 27+6
time till birth | randomisation till birth, maximum 25 weeks
  time span from enrollment to birth
birth weight of neonate | at birth
  birth weight in gram recorded at the hospital
Fetal or neonatal death | at birth, within first 24 hours
  death of the neonate before birth / within first 24 hrs
Need (days) for neonatal special care unit | birth till discharge from hospital, recorded for at least first 48 hrs after birth
  Number of days the neonate is transferred to ICU for medical intervention other than supervision
neonatal morbidity | birth till discharge from hospital, recorded for at least first 48 hrs after birth
  rate of major adverse neonatal outcomes (Intraventricular Haemorrhage III-IV, Retinopathy of prematurity, Respiratory Distress Syndrome II-IV, Need for ventilation > 72 h, Necrotising enterocolitis, Proven or suspected sepsis (antibiotics >5 days)
harm from intervention (neonate) | birth till discharge from hospital, recorded for at least first 48 hrs after birth
  recording any harm of the neonate deriving from the cervical pessary
maternal death | enrollment till discharge from hospital, recorded for at least first 48 hrs after birth
  rate of maternal death due to pregnancy / birth
rate of significant maternal adverse events | enrollment till discharge from hospital, recorded for at least first 48 hrs after birth
  rate of heavy bleeding, cervical tear due to pessary placement, uterine rupture
infection / inflammation | enrollment till discharge from hospital, recorded for at least first 48 hrs after birth
  rate of maternal infection / inflammation during pregnancy / birth
physical or psychological intolerance to cervical pessary | time from placement of cervical pessary at enrollment till removal of cervical pessary at WoG 37, maximum 21 weeks
  rate of maternal physical or psychological intolerance to cervical pessary during pregnancy
hospitalisation for threatened preterm labour before 31 +6 weeks of gestation | enrollment till birth, maximum 21 weeks
  recording of days of hospitalisation for threatened preterm labour before 31 +6 weeks of gestation and recording tocolytic treatment (type/ days/dose)
premature rupture of membranes (ProM) before 31 +6 weeks of gestation | enrollment till birth, maximum 21 weeks
  rate of women with premature rupture of membranes (ProM) before 31 +6 weeks of gestation

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis Kyvernitakis, MD, PhD, Study Director — Buergerhospital Frankfurt
Locations (10):
- University of Adelaide, Adelaide, Australia
- Germany (6):
  - Charite-Universitätsmedizin Berlin, Berlin
  - Vivantes Klinikum im Friedrichshain, Berlin
  - Bürgerhospital Frankfurt/M., Frankfurt
  - Universitätsklinikum Frankfurt, Frankfurt
  - Asklepios Kliniken Krankenhaus Barmbeck, Hamburg
  - Universitätsklinikum des Saarlandes, Homburg
- Greece (2):
  - University Hospital of Athens, Athens
  - Medical School of Aristotle-University of Thessaloniki, Thessaloniki
- Vall d'Hebron University Hospital, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-31): https://cdn.clinicaltrials.gov/large-docs/11/NCT03418311/Prot_SAP_000.pdf